CLINICAL TRIAL: NCT02390505
Title: Role of Vitamin C at 6 Months on Incidence of Complex Regional Pain Syndrome Type I in Upper Limb Surgery
Acronym: SDRC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PI2015_843_0001; 2015-000145-24 (EudraCT Number)
Record Dates: First submitted 2015-02-16; First posted 2015-03-17 (Estimated); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Complex Regional Pain Syndrome (CRPS) TYPE I
Keywords: vitamin C; CRPS; Upper limb surgery
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin C (Experimental): Patients receive vitamin C at a daily dose of 500 mg orally: 7 days before and during 6 weeks after surgery
  Interventions: Drug: Vitamin C
- Placebo (Placebo Comparator): Patients receive placebo at a daily dose of 500 mg orally: 7 days before and during 6 weeks after surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin C
  Arms: Vitamin C
Drug: Placebo
  Arms: Placebo

SUMMARY:
Vitamin C with its antioxidant role has many indications. The objective of this study is to demonstrate that taking vitamin C as a preventive significantly reduces the occurrence of complex regional pain syndrome (CRPS) type 1 in the aftermath of a scheduled surgery of the upper limb.

DETAILED DESCRIPTION:
The preventive role of vitamin C on the development of CRPS type 1 was already demonstrated in traumatology and foot surgery.

The management of CRPS type 1 is long and expensive. A preventive care seems beneficial. Some studies already performed suggest a similar role in scheduled surgery of the upper limb, major provider of CRPS type 1.The aim of the study is to demonstrate a significant reduction of CRPS 1 when taking vitamin C during the perioperative period in upper limb surgery. It is a prospective, randomized, double-blind, with placebo use, in two parallel group, multicenter and national. Patients are followed by their surgeon, under the terms of monitoring their disease. Two visits are required: one at 6 months and at 12 months. The patients will be reviewed at least in the two consultations looking for CRPS type 1 according to the criteria of the International Association for the Study of Pain (IASP)

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 yo
* patients undergoing major surgery of the upper limb
* patients able to give their consent to follow the protocol of treatment and monitoring.

Exclusion Criteria:

* children,
* patients under guardianship,
* pregnant or lactating women,
* patients with hemochromatosis,
* allergy or known hypersensitivity to one of the molecules of treatment,
* patients suffering or having already suffered from complex regional pain syndrome type 1 or type 2,
* patients unable due to personal or professional mobility, to conduct post-operative follow up,
* patients undergoing surgery with nerve suture with nerve graft, emergency surgery,
* patients with glucose-6-phosphate dehydrogenase (G6PD) deficiency,
* patients with chronic kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-07-18 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Appearance of a complex regional pain syndrome (CRPS) 6 months after surgery | 6 months after surgery
  Comparison of the occurrence of participants with CRPS type 1, between the two arms

SECONDARY OUTCOMES:
Appearance of a complex regional pain syndrome 12 months after surgery | 12 months after surgery
  Comparison of the occurrence of participants with CRPS type 1, between the two arms
Tolerance | 6 months after surgery
  Evaluation of tolerance of vitamin C in pre- and post-operative period by adverse events registration
Observance to treatment | 6 months after surgery
  The observance to the treatment is estimated based on an adherence form completed by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel DAVID, MD, Principal Investigator — CHU Amiens
Locations (3):
- France (3):
  - CHU Amiens, Amiens
  - CHU Rouen, Rouen
  - CH Saint-Quentin, Saint-Quentin